CLINICAL TRIAL: NCT02392351
Title: A Boston Scientific Clinical Trial of Renal Denervation Using the Vessix Reduce™ Catheter and Vessix™ Generator for the Treatment of HyperTensioN: REINFORCE
Brief Title: Renal Denervation Using the Vessix Renal Denervation System for the Treatment of Hypertension (REDUCE HTN:REINFORCE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2333
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Renal Denervation (Experimental): Percutaneous renal denervation using the Vessix Reduce™ Catheter and Vessix™ Generator (Vessix Renal Denervation System).
  Interventions: Device: Renal Denervation (Vessix)
- Masked Procedure (Sham Comparator): Percutaneous renal angiography
  Interventions: Device: Renal Angiography

INTERVENTIONS:
Device: Renal Denervation (Vessix) — Percutaneous renal denervation using the Vessix Reduce™ Catheter and Vessix™ Generator
  Other Names: Vessix Reduce™ Catheter and Vessix™ Generator; Vessix Renal Denervation System
  Arms: Renal Denervation
Device: Renal Angiography — Percutaneous renal angiography
  Other Names: Renal Angiogram
  Arms: Masked Procedure

SUMMARY:
The REDUCE HTN: REINFORCE study is being conducted to determine whether the Vessix Reduce™ Catheter and Vessix™ Generator for the treatment of uncontrolled hypertension (off-treatment office systolic blood pressure ≥150 mmHg and ≤180 mmHg) shows acceptable performance at 8 weeks when compared to a masked procedure (renal angiogram).

DETAILED DESCRIPTION:
Prospective, multicenter, single blinded, randomized, controlled, pilot study. Subjects will be randomized to renal denervation treatment or masked renal angiogram procedure (2:1).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years
* OSBP ≥150 mmHg and ≤180 mmHg based on an average of 3 office-based blood pressure measurements
* Average 24-hour ASBP ≥135 mmHg and ≤170 mmHg
* For each kidney, a main renal artery, with or without accessory renal arteries, with diameter ≥3.0 mm and ≤7.0 mm and length ≥20.0 mm
* Agrees to have all study procedures performed, and is competent and willing to provide written, informed consent

Exclusion Criteria:

* Stenosis >30% or renal artery aneurysm in either renal artery
* Fibromuscular dysplasia (FMD)
* Known causes of secondary HTN
* Type 1 diabetes mellitus
* eGFR <40 mL/min/1.73m2
* Known ejection fraction of <30% or heart failure that required hospitalization in the previous 6 months
* Severe valvular heart disease
* ≥1 episode(s) of orthostatic hypotension not related to medication changes (reduction of SBP of ≥20 mmHg or DBP of ≥10 mmHg within three minutes of standing) coupled with symptoms within the past year or during screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09-07 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University; Michael Weber, MD, Principal Investigator — SUNY Downstate College of Medicine
Locations (12):
- United States (12):
  - Cardiology, PC, Birmingham, Alabama
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Cardiovascular Institute of the South, Houma, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Dallas Medical Center, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Aspirus Heart and Vascular Institute, Wausau, Wisconsin

REFERENCES:
- [Derived] Weber MA, Kirtane AJ, Weir MR, Radhakrishnan J, Das T, Berk M, Mendelsohn F, Bouchard A, Larrain G, Haase M, Diaz-Cartelle J, Leon MB. The REDUCE HTN: REINFORCE: Randomized, Sham-Controlled Trial of Bipolar Radiofrequency Renal Denervation for the Treatment of Hypertension. JACC Cardiovasc Interv. 2020 Feb 24;13(4):461-470. doi: 10.1016/j.jcin.2019.10.061. PMID 32081240

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Denervation | Masked Procedure
Started | 34 | 17
Completed | 0 (Primary endpoint: only observational results available.) | 0 (Primary endpoint: only observational results available.)
Not Completed | 34 | 17

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is not different from the assignment in the participant flow. Of note, subjects with multiple ethnic categories are considered independently.
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Denervation | Masked Procedure | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.1) | 58.2 (9.8) | 58.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 20
  Male | 18 | 13 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Caucasian | 27 | 14 | 41
  Hispanic or Latino | 1 | 1 | 2
  Black, of African Heritage | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 34 | 17 | 51
Left Renal Artery [Count of Participants; unit: Participants] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  Participants | 34 | 17 | 51
Left Renal Accessory Artery [Count of Participants; unit: Participants] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  Participants | 5 | 4 | 9
Right Renal Artery [Count of Participants; unit: Participants] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  Participants | 34 | 17 | 51
Right Renal Accessory Artery [Count of Participants; unit: Participants] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  Participants | 5 | 6 | 11
Max Renal Artery Diameter [Mean (Standard Deviation); unit: mm] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  mm | 6.3 (1.3) | 6.1 (1.2) | 6.2 (1.3)
Reference Renal Artery Diameter [Mean (Standard Deviation); unit: mm] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  mm | 5.4 (1.2) | 5.5 (1.1) | 5.5 (1.1)
Renal Artery Length [Mean (Standard Deviation); unit: mm] — Measurements are pre-procedure renal artery characteristics as reported by the core lab.
  mm | 42.0 (17.8) | 46.3 (18.3) | 43.6 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: OBSERVATIONAL: Change (Mean Reduction) in Average 24-hour Ambulatory Systolic Blood Pressure (ASBP) Through 8 Weeks
Description: Change (mean reduction) in average 24-hour Ambulatory Systolic Blood Pressure (ASBP) through 8 weeks post randomization in subjects treated with renal denervation (Test) and subjects treated with masked procedure (Control)
Time Frame: Through 8 weeks
Population: Number analyzed is based upon participants with a complete, valid Ambulatory Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 32 | 15
mmHg | -5.3 (10.1) | -8.5 (9.4)

2. Secondary Outcome: Number of Hospitalizations Due to Severe Hypotension/Syncope
Description: Number of hospitalizations due to severe hypotension/syncope through 6 months.
Time Frame: Through 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

3. Secondary Outcome: Significant Embolic Event Resulting in End-organ Damage or Intervention to Prevent it
Description: Number of subjects experiencing a significant embolic event resulting in end-organ damage or intervention to prevent end-organ damage through 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

4. Secondary Outcome: Renal Artery Dissection or Perforation Requiring Intervention
Description: Number of renal artery dissection or perforation requiring intervention through 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

5. Secondary Outcome: Vascular Complications
Description: Number of vascular complications through 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

6. Secondary Outcome: Significant New Renal Artery Stenosis
Description: Number of significant new renal artery stenosis events through 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

7. Secondary Outcome: Number of Subjects Utilizing Anti-hypertensive Medications
Description: Number of subjects utilizing anti-hypertensive medications at 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 32 | 17
Participants | 16 | 9

8. Secondary Outcome: Mean Reduction in Average 24-hour Ambulatory Systolic Blood Pressure at 6 Months
Description: Change (mean reduction) in the average 24-hour ambulatory systolic blood pressure at 6 months compared to baseline
Time Frame: 6 Months
Population: Number analyzed is based upon participants with a complete, valid Ambulatory Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 30 | 15
mmHg | -16.7 (13.6) | -9.5 (11.4)

9. Secondary Outcome: Mean Reduction in Average 24-hour Ambulatory Diastolic Blood Pressure Through 6 Months
Description: Change (mean reduction) in average 24-hour ambulatory diastolic blood pressure at 6 months compared to baseline.
Time Frame: 6 Months
Population: Number analyzed is based upon participants with a complete, valid Ambulatory Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 30 | 15
mmHg | -9.1 (8.3) | -5.5 (8.2)

10. Secondary Outcome: Number of Subjects Utilizing Anti-hypertensive Medications
Description: Number of subjects utilizing anti-hypertensive medications at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 33 | 17
Participants | 26 | 14

11. Secondary Outcome: Mean Reduction in Average 24-Hour Ambulatory Systolic Blood Pressure
Description: Mean Reduction in Average 24-Hour Ambulatory systolic blood pressure at 12 months
Time Frame: 12 Months
Population: Number analyzed is based upon participants with a complete, valid Ambulatory Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 29 | 12
mmHg | -18.2 (14.3) | -14.3 (8.4)

12. Secondary Outcome: Mean Reduction in Average 24-hour Ambulatory Diastolic Blood Pressure
Description: Mean reduction in average 24-hour ambulatory diastolic blood pressure at 12 months
Time Frame: 12 Months
Population: Number analyzed is based upon participants with a complete, valid Ambulatory Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 29 | 12
mmHg | -11.0 (9.8) | -9.0 (5.7)

13. Secondary Outcome: All-Cause Death
Description: Number of all causes of death through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Renal Failure
Description: Number of renal failure events through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 2 | 0

15. Secondary Outcome: Number of Participants With Hypertensive Crisis
Description: Number of hypertensive crisis events through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 1 | 0

16. Secondary Outcome: Mean Reduction in Average Office-based Systolic Blood Pressure
Description: Mean Reduction in Average office-based systolic blood pressure through 24 months
Time Frame: 24 Months
Population: Number analyzed is based upon participants with a completed Office-Based Systolic Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 30 | 11
mmHg | -19.7 (18.9) | -25.7 (21.2)

17. Secondary Outcome: Mean Reduction in Average Office-based Diastolic Blood Pressure
Description: Mean Reduction in Office-based diastolic blood pressure through 24 months
Time Frame: 24 Months
Population: Number analyzed is based upon participants with a completed Office-Based Systolic Blood Pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 30 | 11
mmHg | -9.5 (10.3) | -9.8 (12.5)

18. Secondary Outcome: Percent of Subjects at Target Blood Pressure
Description: Percent of subjects at target blood pressure through 24 months
Time Frame: 24 Months
Population: Number analyzed is based upon participants with a completed Office-Based Systolic Blood Pressure assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 30 | 11
Participants | 12 | 5

19. Secondary Outcome: Congestive Heart Failure
Description: Number of subjects with congestive heart failure through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 1 | 0

20. Secondary Outcome: Myocardial Infarction
Description: Number of subjects who experience myocardial infarction through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

21. Secondary Outcome: Stroke
Description: Number of subjects experiencing stroke through 24 months
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Masked Procedure
Number analyzed (Participants) | 34 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be collected through 36 months from enrollment.
Description: Enrollment terminated. No endpoint analysis conducted.
Groups:
- Treatment Group: Percutaneous renal denervation using the Vessix Reduce™ Catheter and Vessix™ Generator (Vessix Renal Denervation System)
  Renal Denervation (Vessix): Percutaneous renal denervation using the Vessix Reduce™ Catheter and Vessix™ Generator Through 6 Months
- Masked Procedure - Control Group: Percutaneous renal angiography
  Renal Angiography: Percutaneous renal angiography
Arm/Group | Treatment Group | Masked Procedure - Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 5/34 | 5/17
Other Adverse Events (participants affected / at risk) | 27/34 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=34) | Masked Procedure - Control Group (N=17)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=34) | Masked Procedure - Control Group (N=17)
Hypertension (Vascular disorders) | 11 (13) | 4 (5)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 6 (7)
Dizziness (Nervous system disorders) | 2 (5) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Adverse drug reaction (General disorders) | 4 (7) | 1 (2)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery dissection (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Blood aldosterone increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 1 (1) | 0 (0)
Heart sounds abnormal (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02392351/Prot_SAP_000.pdf